CLINICAL TRIAL: NCT06727864
Title: Safety and Efficacy of Four-month Short Course Regimen in Low Risk Active Tuberculosis- a Multicenter Randomized Controlled Trial
Brief Title: Short Course Regimen in Low Risk Active Tuberculosis- a Multicenter, Randomized, Active-controlled, Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other); Far Eastern Memorial Hospital (Other); E-DA Hospital (Other); Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Susan Shin-Jung Lee, Attending physician, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSVGH24-CT2-16
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Tuberculosis
Keywords: tuberculosis; short course regimen; safety; sputum conversion; recurrence rate
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: Two months of isoniazid (H), pyrazinamide (Z), rifampicin (R), and pyrazinamide (Z) Subsequent orders are for H(E)Z for another two months
Masking Description: Masking will not be done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention/Treatment (Experimental): Two months of isoniazid (H), ethambutol (E), rifampicin (R) and Pyrazinamide (Z) followed by HR(E) for another two months
  Interventions: Drug: 4-month regimen (2HERZ/2HRE)
- 6-months HERZ (2HERZ/4HRE) (Active Comparator): Two months of isoniazid (H), pyrazinamide (Z), rifampicin (R) and Pyrazinamide (Z) followed by HR(E) for another four months
  Interventions: Drug: 6-month (2HERZ/4HRE)

INTERVENTIONS:
Drug: 4-month regimen (2HERZ/2HRE) — 4-month (2HERZ/2HRE)
  Arms: Intervention/Treatment
Drug: 6-month (2HERZ/4HRE) — 2 months of HREZ followed by 4 months of HR/HRE
  Arms: 6-months HERZ (2HERZ/4HRE)

SUMMARY:
Tuberculosis remains an important global health problem, and the world is currently not on track to end the TB epidemic by 2030. With the concerted efforts of the government and medical community, the incidence of TB in Taiwan has gradually decreased, however, Taiwan remains an endemic area for TB. The development of efficacious, safe, and shorter treatment regimens could significantly improve treatment completion rate and reduce transmission of TB. The current treatment guidelines for drug-susceptible TB from the World Health Organization (WHO), American Thoracic Society (ATS), United States Center for Diseases Control (U.S. CDC), Infectious Diseases Society of America (IDSA) and European Respiratory Society (ERS) include 2 months of isoniazid, rifampin, pyrazinamide and ethambutol (HREZ), followed by 4 months of isoniazid, rifampin, and ethambutol(HRE). The current treatment regimen requires 6 months of treatment, despite being highly efficacious, requires long duration of treatment. Adherence to treatment is the major barrier which poses a negative impact to TB control, and increased cost to both the patient and the public health system. Developing an efficacious, safe and short treatment regimen can significantly improve TB management and treatment success rates.

DETAILED DESCRIPTION:
This prospective, multicenter, randomized, open-labeled 3-year study, will recruit 270 adult patients with newly diagnosed tuberculosis with low risk of recurrence, and randomized 1:1 to a 4 months 2HREZ/2HRE (n=135) versus standard, 6 months regimen 2HREZ/4HRE (n=135). Expected enrollment will be 90 patients in year 1, 90 in year 2 and 90 in year 3.

This study aims to evaluate the efficacy, safety and long-term recurrence rate of a short-course, 4-months regimen including 2HREZ/2HRE compared with the standard 6-months regimen, 2HREZ/4HRE, and the impact of short regimen on reducing the costs and loading to the public health and medical system

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed pulmonary tuberculosis patients combined with any of the following diagnostic conditions:

  * at least one set of sputum specimens is positive for Mycobacterium tuberculosis culture or TB PCR test; or
  * pathological and histological findings of typical tuberculosis manifestations;
  * clinical diagnosis and Physician determines the need for complete anti-tuberculosis treatment
* Those who have had tuberculosis in the past and have been cured for at least three years can be included
* Aged over 20 years old
* Laboratory data at the time of inclusion in the study or within 14 days:

  * Serum or plasma glutamic acid pyruvate transaminase (ALT) value ≦ three times the upper limit of normal
  * Serum or plasma total bilirubin ≦ 2.5 times the upper limit of normal
  * Serum or plasma creatinine ≦ twice the upper limit of normal or creatinine clearance greater than 30 mL/min
  * Heme ≧7.0 g/Dl
  * Platelets ≧100,000/mm3
* Patient signs consent form
* Patients who agree to join and cooperate with the county and city health bureau's urban treatment plan to ensure medication compliance.

Exclusion Criteria:

* The acid-fast smear of sputum or respiratory specimen is strongly positive (≥ 2+)
* Chest X-ray or lung computed tomography combined with open lesions
* Chest X-ray or lung computed tomography shows extensive lesions and the clinician judges that short-term treatment is not suitable
* Simultaneous combination of intrapulmonary and extrapulmonary tuberculosis
* People who are unable to take oral medications
* People who have participated in this research
* Have used anti-tuberculosis drugs for more than 14 days
* A history of tuberculosis suspected or diagnosed as central nervous system tuberculosis, bone or joint tuberculosis, miliary tuberculosis or tuberculous pericarditis.
* Known history of allergy or intolerance to this study drug
* Patients with HIV infection, organ transplantation, and chronic renal failure
* Long-term use of immunosuppressive drugs, including steroid use >10mg/day (more than 30 consecutive days in the last three months)
* Late exclusion: Mycobacterium tuberculosis is known to be resistant to any one or more of the following drugs: rifampin, isoniazid, ethambutol

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
TB disease free survival at 12 months post-randomization | 12 months
  Number of participants without TB disease at 12 months after randomization
TB disease free survival at 24 months post randomization | 24 months
  Number of participants without TB disease at 24 months after randomization
Grade 3-5 adverse events | From enrollment to the end of treatment at 4 or 6 months
  Development of Grade3-5 adverse events during treatment

SECONDARY OUTCOMES:
Early sterilizing activity | 8 weeks
  The proportion of patients with a negative sputum culture at the end of intensive phase therapy at 8 weeks
Sputum culture conversion | 4, 8, 12, 16,20,24 weeks,3, 6, 12 and 24 months after treatment
  Time to stable sputum culture conversion
All-cause mortality | 4, 12 months
  All-cause mortality at 4 months and 12 months post-treatment assignment
Attributable mortality | 4, 12 months
  Attributable mortality at 4 months and 12 months post-treatment assignment
Changes in interferon-gamma levels | 2, 4, 8, 12,16or 24 weeks
  Changes in interferon-gamma levels during treatment compared to baseline
Changes in tumor necrosis factor-alpha levels | 2, 4, 8, 12,16or 24 weeks
  Changes in tumor necrosis factor-alpha levels during treatment compared to baseline
Changes in interleukin-12 and interleukin-6 levels | 2, 4, 8, 12,16or 24 weeks
  Changes in interleukin-12 and interleukin-6 levels during treatment compared to baseline
Changes in triggering receptor expressed on myeloid cells-1 (TREM-1) levels | 2, 4, 8, 12,16or 24 weeks
  Changes in triggering receptor expressed on myeloid cells-1 (TREM-1) levels during treatment compared to baseline

OTHER OUTCOMES:
HLA associations with severe drug adverse events | Upon joining or within two weeks of study entry
  HLA Genotyping to detect predictors for occurrence of severe drug adverse events including skin rash and hepatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shin-Jung Lee, MD, PhD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (8):
- Taiwan (8):
  - Far Eastern Memorial Hospital, New Taipei City, Bangiao
  - Taichung Hospital, Taichung, West
  - E-DA Healthcare Group, Kaoshiung, Yanchao
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: Undecided